CLINICAL TRIAL: NCT07201883
Title: A Randomized Clinical Trial; Chewing Gum vs. Ondansetron as Rescue Treatment for PONV in Female Patients Undergoing Laparoscopic Surgery at a Single Centre in Lebanon
Brief Title: Chewing Gum vs. Ondansetron as Rescue Treatment for PONV in Female Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Omar Rajab, Chairman of Anesthesia Department, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MGH-07-25038
Record Dates: First submitted 2025-08-22; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Nausea and Vomiting (PONV)
Keywords: PONV; Ondansetron; Postoperative Period; Vomiting; Laparoscopy; Antiemetics
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Ondansetron; Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ondansetron (Active Comparator)
  Interventions: Drug: Ondansetron (Zofran)
- Chewing Gum (Experimental)
  Interventions: Other: chewing gum
- Ondansetron + Chewing Gum (Sham Comparator)
  Interventions: Combination Product: Ondansetron + Chewing gum

INTERVENTIONS:
Drug: Ondansetron (Zofran) — 4 mg IV push
  Arms: Ondansetron
Other: chewing gum — Peppermint sugar free chewing gum
  Arms: Chewing Gum
Combination Product: Ondansetron + Chewing gum — Ondansetron 4 mg IV push Peppermint sugar free chewing gum
  Arms: Ondansetron + Chewing Gum

SUMMARY:
The proposed randomized clinical trial aims to test and compare the efficacy of chewing gum vs. Intravenous antiemetic ondansetron as rescue treatment for post-operative nausea and vomiting (PONV) among Lebanese female patients undergoing laparoscopic surgery in the post-operative anesthesia care unit (PACU).

DETAILED DESCRIPTION:
Post-operative nausea and vomiting remains a significant complication following general anesthesia, particularly when volatile anesthetics are used. Previous studies, including a multicenter randomized trial conducted in Australia, have explored alternative treatment modalities for PONV. Chewing gum, a non-pharmacological intervention, has shown promise as a potential alternative or adjunct to conventional antiemetics like ondansetron. This study focuses on the Lebanese female population, aged 18 and above, who have undergone laparoscopic surgery under volatile anesthetic-based general anesthesia. This demographic is chosen based on established risk factors for PONV and may offer unique insights into efficacy within this subgroup.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Aged 18 and above,
* Weight 40kg and above,
* Who have undergone laparoscopic
* Surgery under volatile anesthetic-based general anesthesia.

Exclusion Criteria:

* Have history of motion sickness,
* Maintained anesthesia during surgery using Propofol-pump
* Were given antiemetics within 8 hours pre-surgery
* Allergy to ondansetron
* Planned mechanical ventilation post-operation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Complete cessation of PONV with no recurrence and no rescue medication | 2 hours

SECONDARY OUTCOMES:
Patient satisfaction | post-operative period ( up to 3 hours)
Quantity of rescue treatment modalities used | immediately after PONV start until complete resolution of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Makassed General Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chernik DA, Gillings D, Laine H, Hendler J, Silver JM, Davidson AB, Schwam EM, Siegel JL. Validity and reliability of the Observer's Assessment of Alertness/Sedation Scale: study with intravenous midazolam. J Clin Psychopharmacol. 1990 Aug;10(4):244-51. PMID 2286697
- See also: Related Info — https://journals.lww.com/lww-medicalcare/abstract/1996/03000/a_12_item_short_form_health_survey__construction.3.aspx